CLINICAL TRIAL: NCT03148977
Title: Evaluating a Point-of-Care, Quantitative Matrix Metalloproteinase Assay as a Predictor of Successful Graft Take in Patients Undergoing Cutaneous Auto Grafting for Acute Burn Injury- A Pilot Study
Brief Title: Evaluating MMPs in Burns
Status: Terminated | Type: Observational
Why Stopped: IRB expired
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201602508
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Burns; Thermal Burn; Thermal Injury
Keywords: Matrix Metalloproteinases
MeSH Terms: conditions — Burns | interventions — Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Acute burn wound exudate Acute burn wound tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to the burn center: Patients admitted to the Burn Service with acute burn injuries requiring at least one surgical excision and grafting operation.
  Interventions: Procedure: Graft

INTERVENTIONS:
Procedure: Graft — Autogenous skin grafting is the only definitive treatment for the full thickness burn injuries, and thus represents the centerpiece of modern burn care.

SUMMARY:
The objective of this study is to determine whether our chemical assay can be used to reliably predict graft take or failure in patients undergoing autologous skin grafting for treatment of acute burn injury.

DETAILED DESCRIPTION:
This is an observational pilot study of patients treated at UF Health Shands Burn Center adult service. This is a study to determine the predictive value of quantifying concentrations of specific MMPs. Coupling this with a specialized collection sample collection system and a calibrated fluorimetry allows for the rapid assessment of MMP concentrations. This assay has been validated as a predictor of failed wound healing in a published clinical study involving chronic open wounds.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Admitted with acute burns injuries (flame, contact or scald) requiring at least one surgical excision and grafting operation will be considered for inclusion
* Burn injury less than one week old

Exclusion Criteria:

* Electrical, chemical or cold-induced burn injury
* Total body surface area burn >50 %
* Pre injury diagnosis of chronic renal insufficiency, liver failure, refusal to accept blood transfusion or withdrawal of care within three days of admission will also be exclusion criteria
* Patients not expected to survive
* Patients presenting with re-injury to previously burned and treated areas.
* Patients who present after receiving burn excision surgery out an outside facility for the current acute injury

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult burn patients admitted
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Predictability of graft take | 2 years
  Determine whether chemical assay can be used to reliably predict graft take or failure in patients undergoing autologous skin grafting for treatment of acute burn injury.

SECONDARY OUTCOMES:
Wound healing | 2 years
  Assess the predictive value of serial MMP assays in identifying wounds transitioning from likely-to-fail to likely-to-succeed

CONTACTS AND LOCATIONS:
Overall Officials: Joshua S. Carson, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health Cancer Hospital, Gainesville, Florida
  - UF Health Shands at the University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weigelt MA, Lev-Tov HA, Tomic-Canic M, Lee WD, Williams R, Strasfeld D, Kirsner RS, Herman IM. Advanced Wound Diagnostics: Toward Transforming Wound Care into Precision Medicine. Adv Wound Care (New Rochelle). 2022 Jun;11(6):330-359. doi: 10.1089/wound.2020.1319. Epub 2021 Jul 21. PMID 34128387